CLINICAL TRIAL: NCT01119482
Title: The Impact of Vaccination With a Serogroup A Meningococcal Conjugate Vaccine on Carriage of Serogroup A Meningococci in Mali and Niger
Brief Title: Study on the Impact of Vaccination With a Conjugate Vaccine on Meningococcal Carriage
Acronym: MenAfriCar
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: London School of Hygiene and Tropical Medicine (Other)
Collaborators: Bill and Melinda Gates Foundation (Other); Wellcome Trust (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: LSHTM_5698
Record Dates: First submitted 2010-04-21; First posted 2010-05-07 (Estimated); Last update posted 2013-04-19 (Estimated); Status verified 2013-04

CONDITIONS: Meningitis
Keywords: Serogroup A meningococcal vaccine; meningococcal carriage; incidence; prevalence
MeSH Terms: conditions — Meningitis | interventions — MenAfriVac

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Vaccination (Other): Healthy volunteers before and after vaccination
  Interventions: Biological: MenAfriVac™

INTERVENTIONS:
Biological: MenAfriVac™ — Children, adolescents and adults aged 1 to 29 years old will receive a single intramuscular injection of the meningococcal serogroup A conjugate vaccine .
  Other Names: Meningococcal serogroup A conjugate vaccine

SUMMARY:
Meningococcal disease occurs throughout the world but attack rates in the Sahelian and sub-Sahelian regions of Africa - the African meningitis belt - are many times higher than those seen in any other part of the world. During 2009, over 70,000 meningitis cases and 3,200 deaths were reported in Nigeria, Niger, and Chad alone.

In 2001, a public private partnership between WHO and PATH was created, the Meningitis Vaccine Project (MVP). The MVP set out to develop an affordable meningococcal serogroup A conjugate vaccine (MenAfriVac™) for use in the African meningitis belt. This was successfully achieved, and the new vaccine, produced by the Serum Institute of India (SII), was granted a licence in 2009 for international export. The vaccine dossier was submitted to WHO for prequalification at the beginning of 2010. Introduction through mass vaccination is planned in three African Meningitis belt countries in 2010 (Burkina Faso, Mali and Niger). The implementation of MenAfriVac will be the responsibility of the local Ministry of Health, with the support of the World Health Organization.

It is anticipated that this vaccine will be deployed in other countries of the meningitis belt in 2011. This vaccine should provide high levels of direct protection to immunised individuals but, as for serogroup C conjugate vaccines in the United Kingdom, a greater public health impact will be achieved if carriage and transmission of the infection are also prevented.

The London School of Hygiene & Tropical Medicine (LSTHM) is coordinating the African Meningococcal Carriage Consortium (MenAfriCar). One of the primary objectives of the MenAfriCar project is to evaluate the impact of the new conjugate vaccine on meningococcal carriage and transmission of serogroup A meningococci in Mali, Niger and Chad. A community-based prospective, pre- and post intervention, observational study will be conducted. MenAfriCar will also help to develop research capacity in the participating African countries.

DETAILED DESCRIPTION:
Epidemiological information will be obtained at community, household and individual levels.

In each country, informed consent will be obtained from adults selected to participate in the study and for the children under their care. Written informed assent will also be obtained from participants aged 12 to 15 years. Oral assent will be obtained from younger children. Once consent or assent has been obtained, a structured questionnaire will be completed following discussions with the head of the household which records information about sleeping and cooking arrangements in the household. Each study participant or their guardian will complete a questionnaire which collects information on potential risk factors for meningococcal carriage such as occupation, smoking, recent travel, including travel on the pilgrimage, attendance at social gatherings, and recent respiratory infection. Following interview, a pharyngeal swab will be obtained from each study participant. A 5 ml blood sample will be obtained from 200 randomly selected subjects in each of the four older age categories and from 50 infants aged 6 - 11 months (a total of 850 samples) during the initial survey to measure serogroup A bactericidal and Immunoglobulin G ELISA serogroup A, C, W135, X and Y meningococcal antibodies. Blood will not be collected from infants under the age of 6 months.

In each country, immediate processing of pharyngeal swabs will allow the identification of subjects who are carrying meningococci and the serogroup of these meningococci will be determined within 2 - 4 days of collection of the sample. The households of these subjects will be visited as soon as possible after identification of a carrier has been made, informed consent will be obtained and if the participant agrees, a pharyngeal swab will be obtained twice a month for two months and monthly for a further four months, a total of 8 follow-up samples to estimate the rates of acquisition and loss of carriage in household's contacts. During the first visit, a 5 ml blood sample will be obtained from all subjects over the age of 6 months for measurement of IgG ELISA and bactericidal serogroup A meningococcal antibodies to determine concentrations that protect against acquisition of carriage. No further blood samples will be collected. A rapid diagnostic test for malaria will be performed on any subject who is febrile or unwell and antimalarial treatment provided according to the national guidelines if it is positive. The results of these household studies will show the impact of vaccination on acquisition rates of carriage.

Similar cross-sectional and longitudinal surveys to those described above will be conducted approximately 6 and 18 months after the mass vaccination campaigns with the serogroup A meningococcal conjugate vaccine.

AMENDMENT TO ORIGINAL STUDY PROTOCOL:

The initial proposal included provision for an interview to collect information on potential risk factors for carriage, collection of a pharyngeal swab from each study participant, and 8 swabs from household contacts of index carriers over a six-month period. It included provision for the collection of one 5 ml blood sample during the initial cross-sectional survey from 800 subjects aged 6 months or older for baseline serological assays, and for collection of a further 5 ml post-vaccination sample. It also included provision for collection of a 5 ml blood sample from all subjects over the age of 6 months during the first visit of the household follow up study to determine concentrations that protect against acquisition of carriage.

During pre-vaccination surveys conducted in 2010, pharyngeal swabs were collected from 4,300 and 5,000 age stratified subjects in Mali and Niger respectively. Molecular analysis performed in Oxford, confirmed that there was no serogroup A meningococci among the 48 and 338 isolates of putative meningococci identified in Mali and Niger respectively. In contrast, serogroup A meningococcal carriers were identified in Chad during the course of a related epidemiological study (REF.5699). In addition, during the 2011 African meningitis season, more than 90% of cases of serogroup A meningococcal disease recorded in the meningitis belt came from Chad or Cameroun with very few cases being reported from Mali or Niger. These observations indicate that it may be possible to measure the impact of MenAfriVac™ on serogroup A meningococcal in Chad rather than in Mali or Niger as had been proposed originally.

For the reasons indicated above, it is proposed to undertake a pre-vaccination carriage survey in Chad in 5,000 subjects in the 2011 rainy season instead of the 2,000 subjects proposed originally for the epidemiological study (REF. 5698). As the prevalence of carriage was higher in rural than in urban areas in the 2010 rainy season surveys conducted in Chad, we propose to study 4000 subjects in two rural areas and 1,000 subjects in an urban area. This will allow a comparison to be made with the results obtained in the 2010 rainy season survey when 1000 subjects were recruited in urban and rural areas respectively.

The same study procedures described in original proposal will be performed in Chad, except that no blood samples will be obtained during the initial survey as these were collected during 2010. However, one blood sample will be obtained from household contacts of index carriers as set out for the surveys originally planned for Mali and Niger. The same consent form as the one proposed initially will be used.

Depending upon the prevalence of serogroup A meningococcal carriage in the 2011 rainy season survey conducted in Chad, a decision will be made as to whether or not to proceed with two post-vaccination surveys as indicated in the original protocol for Mali and Niger. Vaccination of the whole of Chad with MenAfriVac™ will commence in the last quarter of 2011 and the whole country is likely to be covered by early 2012.

ELIGIBILITY:
Inclusion Criteria:

* Adults or children whose parent or guardian give consent to participate in the study
* Adults or children who do not have a serious acute or chronic illness

Exclusion Criteria:

* lack of consent given by an adult or the parent or guardian of a potentially eligible study child
* Adults or children who have a serious acute or chronic illness

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 33000 (Actual)
Dates: Start 2010-05; Primary Completion 2012-05 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
Meningococcal carriage | Prevalence of meningococcal carriage at six months after vaccination
  Cross-sectional surveys will be conducted in approximately 5,000 age stratified subjects before and 6 and 18 months after vaccination with the meningococcal serogroup A conjugate vaccine to estimate the prevalence of meningococcal carriage. During each cross-sectional survey all household members in contact with an identified serogroup A carrier will be included in a household follow up study to investigate the impact of vaccination on the rates of acquisition of meningococcal carriage.

SECONDARY OUTCOMES:
Meningococcal carriage | Prevalence of meningococcal carriage at 18 months after vaccination
  Cross-sectional surveys will be conducted in approximately 5,000 age stratified subjects before and 6 and 18 months after vaccination with the meningococcal serogroup A conjugate vaccine to estimate the prevalence of meningococcal carriage. During each cross-sectional survey all household members in contact with an identified serogroup A carrier will be included in a household follow up study to investigate the impact of vaccination on the rates of acquisition of meningococcal carriage.

CONTACTS AND LOCATIONS:
Overall Officials: Maria C Nascimento, MD, PhD, Study Director — London School of Hygiene and Tropical Medicine; Brian Greenwood, MD, Principal Investigator — London School of Hygiene and Tropical Medicine
Locations (3):
- Centre de Support en Sante Internationale (CSSI), Ndjanema, Chad
- Center for Vaccine Development, Mali, Bamako, Bamako, Mali
- Centre de Recherche Médicale et Sanitaire, Niamey, Niger

REFERENCES:
- [Derived] Diallo K, Gamougam K, Daugla DM, Harrison OB, Bray JE, Caugant DA, Lucidarme J, Trotter CL, Hassan-King M, Stuart JM, Manigart O, Greenwood BM, Maiden MCJ. Hierarchical genomic analysis of carried and invasive serogroup A Neisseria meningitidis during the 2011 epidemic in Chad. BMC Genomics. 2017 May 22;18(1):398. doi: 10.1186/s12864-017-3789-0. PMID 28532434